CLINICAL TRIAL: NCT03517709
Title: Feasibility of Home Telehealth Monitoring for Improvement in Management of Hypertension for Secondary Stroke Prevention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No recruitment of subjects
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00119776
Record Dates: First submitted 2017-12-18; First posted 2018-05-07 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Stroke; Hypertension
MeSH Terms: conditions — Stroke; Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Conventional (Other)
  Interventions: Other: Primary Care Physician Management of blood pressure
- Blood Pressure Monitor (Other)
  Interventions: Device: Withings Smart Blood Pressure Monitor

INTERVENTIONS:
Other: Primary Care Physician Management of blood pressure — * You will receive a 30-minute education session about your blood pressure medications and the need to take them every day.
  * Your primary care physician will make recommendations on your optimal target blood pressure range and medication recommendations. .
  Arms: Conventional
Device: Withings Smart Blood Pressure Monitor — We will use the Withings Smart Blood Pressure Monitor for daily blood pressure measurements.
  Arms: Blood Pressure Monitor

SUMMARY:
This research is being done to determine how home blood pressure monitoring, using a commercially available blood pressure monitor with the capability of transmitting readings to stroke doctors can help manage blood pressure in the optimal range after a stroke. High blood pressure is the leading risk factor for stroke. It is important to control high blood pressure after a stroke to prevent another one from happening. We will use the Withings Smart Blood Pressure Monitor for daily blood pressure measurements.

Tracking of blood pressure measurements will be done via iPod Touch equipped with internet connectivity. We hope to learn if this method of managing blood pressure is more effective than the standard way of having patients visit primary care physicians (the control group for this study). We will also get feedback from participants who will receive the Withings Smart Blood Pressure Monitor about the ease of use and overall satisfaction with this blood pressure device. People 18-100 years old who have had a stroke in the past 6 months may join. You will be excluded from the study if you are pregnant or plan on becoming pregnant in the near future.

ELIGIBILITY:
Inclusion Criteria:

* People 18-100 years old who have had a stroke in the past 6 months may join.

Exclusion Criteria:

* You will be excluded from the study if you are pregnant or plan on becoming pregnant in the near future.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 3 months
  The blood pressure will be obtained on Day 90 by measuring three consecutive times and obtaining an average.
Stroke in 90 days | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided